CLINICAL TRIAL: NCT05644860
Title: Nano Composites and Light Cure Composites - A Comparative Assessment of Bond Failure Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2022/19
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Nanotechnology, Dental Materials, Composites
MeSH Terms: interventions — Filtek Z250; Transbond XT

STUDY DESIGN:
Intervention Model Description: The patients meeting the slection criteria chall be randomly allocated in two groups (A and B)/ Brackets in the group A shall be bonded with the conventional composite (Transbond XT, 3M Unitek, USA) with appreciably good shear bond strength. In patients belonging to group B, brackets shall be bonded with nanohybrid composite (Filtek Z250).
  Long term succes shall be evaluated by comparing the bracket failute rate between the two groups.
Who Masked: Participant
Masking Description: The two materials being compared look similar and according to the manufacturers' instructions they are applied using a similar protocol i.e. enamel conditioning, application of unfilled resin, placement of brackets and light curing. Hence the patient will not be able to identify as to which experimental group they are placed in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Composite Group (Transbond XT) (Active Comparator): Patients in which brackets will be bonded with conventional composite resin (Transbond XT)
  Interventions: Combination Product: Conventional Composite Group (Transbond XT)
- Nanohybrid Compisite Group (Filtek Z250) (Experimental): Patients in which brackets will be bonded with nanohybrid composite resin (Filtek Z250)
  Interventions: Combination Product: Nanohybrid Compisite Group (Filtek Z250)

INTERVENTIONS:
Combination Product: Nanohybrid Compisite Group (Filtek Z250) — Orthodontic brackets shall be bonded with Nano hybrid composite
  Arms: Nanohybrid Compisite Group (Filtek Z250)
Combination Product: Conventional Composite Group (Transbond XT) — Patients in which brackets will be bonded with conventional composite resin (Transbond XT)
  Arms: Conventional Composite Group (Transbond XT)

SUMMARY:
This randomized clinical trial is aimed to evaluate the bond failure rates of the brackets bonded with nano-hybrid composites (Filtek Z250) to that of conventional composites (Transbond XT)

DETAILED DESCRIPTION:
Orthodontic brackets are attached to the teeth with a robust bonding material called composite resin, however sometimes the bond between the braket and the tooth surface may fail halting the desired tooth movement. Repeated bond failures like these are inconvenience both for the orthodontists as well as the patients. With each bracket loosening due to bond failure, treatment time is prolonged as the activation planned on eash visit is delayed resuling in increased treatment time.

Nanotechnology has recently made a breakthrough in dental materials through incorporation of nanoparticles. Composites containing nano-filler particles exhibit higher compression strength, flexural strength, elastic modulus and wear resistance (Rabia and Bilal). In vitro studies have shown that nanohbrid composites have shear bond stregnths similar to that of conventional composites however the environment of oral cavity is challenging and there are no long term clinical trials to validate these results.

The aim of this study is to compare the rate of bond failure between the brackets bonded with nano hybrid composites and that of the conventional composites over a period of six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients having treatment with fixed metallic orthodontic appliances
* Patients in whom both upper and lower arches are bonded in single visit

Exclusion Criteria:

* Patients with variations in morphology of teeth
* Patients with defective enamel, dentine and cementum
* Patiens with parafunctioal habits
* Patients with restorations involving the facial surface of teeth

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Bracket failure rate | 6 months
  Number of brackets detached from the tooth surface

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Islamabad/ Federal, Pakistan